CLINICAL TRIAL: NCT07404605
Title: Electrochemotherapy Induces Changes in Tumor Microenvironment of Cutaneous and Subcutaneous Metastases in Patients With Cutaneous Melanoma
Brief Title: Electrochemotherapy-Induced Changes in Tumor Microenvironment in Cutaneous Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OI-EKT-MEL-2023; 0120-297/2023/3 (Other: KME Slovenia)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Skin Cancer; Subcutaneous Metastases
Keywords: electrochemotherapy
MeSH Terms: conditions — Skin Neoplasms | interventions — Electrochemotherapy

STUDY DESIGN:
Intervention Model Description: Single-arm prospective interventional study evaluating tumor microenvironment changes in melanoma metastases before and after electrochemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrochemotherapy (ECT) (Experimental): Patients with cutaneous melanoma with cutaneous and/or subcutaneous metastases undergoing electrochemotherapy as part of clinical management. Electrochemotherapy is performed using intravenous bleomycin or intratumoral cisplatin. Tumor samples are collected before and after treatment for analysis of tumor microenvironment changes.
  Interventions: Procedure: Electrochemotherapy

INTERVENTIONS:
Procedure: Electrochemotherapy — Electrochemotherapy is performed according to standard clinical procedures with application of electric pulses combined with administration of cytotoxic agents (intravenous bleomycin or intratumoral cisplatin) for treatment of cutaneous and subcutaneous melanoma metastases.

SUMMARY:
Cutaneous melanoma frequently develops cutaneous and subcutaneous metastases, which may cause significant morbidity and negatively affect quality of life. Electrochemotherapy (ECT) is an established local treatment modality for cutaneous and subcutaneous tumor lesions that combines the administration of cytotoxic drugs with the application of electric pulses to increase drug uptake into tumor cells.

In addition to its direct cytotoxic effects, electrochemotherapy may induce changes in the tumor microenvironment, including immune cell infiltration, vascular alterations, and other biological responses that could influence tumor control.

The aim of this study is to evaluate changes in the tumor microenvironment of cutaneous and subcutaneous melanoma metastases following electrochemotherapy with either intravenous bleomycin or intratumoral cisplatin. Tumor tissue samples collected before and after treatment will be analyzed to characterize microenvironmental changes and to compare treated and untreated lesions.

The results of this study may improve understanding of biological effects of electrochemotherapy in melanoma metastases and support further development of treatment strategies.

DETAILED DESCRIPTION:
This is a prospective interventional clinical study designed to investigate electrochemotherapy-induced changes in the tumor microenvironment of cutaneous and subcutaneous melanoma metastases.

Electrochemotherapy is a local treatment approach that combines electroporation with cytotoxic agents in order to increase intracellular drug delivery and enhance tumor cell death. The treatment is routinely used for superficial tumor lesions, including melanoma metastases, and can be performed using intravenous bleomycin or intratumoral cisplatin.

The primary objective of this study is to characterize changes in the tumor microenvironment in melanoma metastases following electrochemotherapy. Tumor tissue samples will be collected from untreated lesions and from lesions treated with electrochemotherapy. Histopathological and immunohistochemical analyses will be performed to evaluate changes in the tumor microenvironment, including cellular and stromal components, immune-related features, and other relevant biological markers.

The study will include patients with cutaneous melanoma presenting with cutaneous and/or subcutaneous metastases who are eligible for electrochemotherapy as part of their clinical management. Electrochemotherapy will be performed according to established clinical procedures using intravenous bleomycin or intratumoral cisplatin. Biopsy or surgical samples will be collected before and after treatment to enable comparative analyses of treated and untreated tumor tissue.

Collected clinical and pathological data will be used to assess associations between treatment-related microenvironmental changes and patient and lesion characteristics. The study aims to provide additional insight into biological effects of electrochemotherapy beyond local tumor control and may contribute to improved understanding of mechanisms involved in treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Histologically confirmed cutaneous melanoma
* Presence of cutaneous and/or subcutaneous metastases eligible for electrochemotherapy
* Candidate for electrochemotherapy with intravenous bleomycin or intratumoral cisplatin according to standard clinical practice
* Ability to provide written informed consent

Exclusion Criteria:

* Contraindication to electrochemotherapy or study drugs (bleomycin or cisplatin)
* Pregnancy or breastfeeding
* Severe comorbidities preventing electrochemotherapy
* Inability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor Microenvironment Markers After Electrochemotherapy | Baseline (pre-treatment) and post-treatment (up to 3 months after electrochemotherapy)
  Comparison of histopathological and immunohistochemical tumor microenvironment characteristics in cutaneous/subcutaneous melanoma metastases before and after electrochemotherapy, including immune cell infiltration and other predefined microenvironmental markers.

SECONDARY OUTCOMES:
Difference in Tumor Microenvironment Between Treated and Untreated Lesions | Up to 3 months after electrochemotherapy
  Comparison of tumor microenvironment markers between electrochemotherapy-treated lesions and untreated lesions in the same patient.
Local Tumor Control of Treated Lesions | Up to 12 months after electrochemotherapy
  Evaluation of local response of treated cutaneous and subcutaneous melanoma metastases after electrochemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No